CLINICAL TRIAL: NCT01164163
Title: A Phase I Study of JAK Inhibition (INCB018424) in Children With Relapsed or Refractory Solid Tumors, Leukemias, and Myeloproliferative Neoplasms
Brief Title: INCB18424 in Treating Young Patients With Relapsed or Refractory Solid Tumor, Leukemia, or Myeloproliferative Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL1011; COG-ADVL1011 (Other: Children's Oncology Group)
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; refractory chronic lymphocytic leukemia; relapsing chronic myelogenous leukemia; childhood myelodysplastic syndromes; previously treated myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; chronic myelomonocytic leukemia; juvenile myelomonocytic leukemia; myelodysplastic/myeloproliferative neoplasm, unclassifiable; polycythemia vera; essential thrombocythemia; childhood acute promyelocytic leukemia (M3); acute myeloid leukemia/transient myeloproliferative disorder; primary myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Leukemia, Myelomonocytic, Juvenile; Polycythemia Vera; Thrombocythemia, Essential; Leukemia, Myeloid, Acute; Myeloproliferative Syndrome, Transient; Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Ruxolitinib) (Experimental)
  Interventions: Drug: ruxolitinib phosphate; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: ruxolitinib phosphate
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: INCB18424 (Ruxolitinib) may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase 1 clinical trial is studying the side effects and best dose of INCB18424 in treating young patients with relapsed or refractory solid tumor, leukemia, or myeloproliferative disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the maximum-tolerated dose and/or recommended phase II dose of oral JAK inhibitor INCB18424 administered continuously, twice daily to pediatric patients with relapsed or refractory solid tumors.
* To define and describe the toxicities of this treatment administered on this schedule in pediatric patients with relapsed or refractory solid tumors, leukemias, or myeloproliferative neoplasms (MPNs).
* To characterize the pharmacokinetics of this treatment in pediatric patients with relapsed or refractory solid tumors, leukemias, or MPNs.

Secondary

* To preliminarily define the antitumor activity of this treatment within the confines of a phase I study.
* To assess the biologic activity of oral JAK inhibitor INCB18424 upon JAK-STAT signaling in pediatric patients with relapsed or refractory solid tumors, leukemias, or MPNs.
* To assess the cytotoxicity and biologic activity of oral JAK inhibitor INCB18424 upon phosphosignaling and mutation burden in pediatric patients whose leukemias or MPNs have known CRLF2 and/or JAK mutations.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive oral JAK inhibitor INCB18424 twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients with relapsed or refractory leukemia may receive intrathecal chemotherapy in course 2 and subsequent courses at the discretion of the treating physician.

Plasma, bone marrow, and blood samples may be collected at baseline, during course 1, and before subsequent courses for pharmacokinetic analysis and correlative biology studies.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of one of the following:

  * Relapsed or refractory extracranial solid tumor
  * Relapsed or refractory leukemia

    * At least 25% blasts in the bone marrow (M3) with the exception of patients with acute myeloid leukemia (AML), who must have > 20% blasts in the bone marrow
  * Relapsed or refractory myeloproliferative neoplasm (MPN)

    * At original diagnosis or relapse
    * Current diagnostic criteria for MPNs include polycythemia vera, essential thrombocythemia, juvenile myelomonocytic leukemia, myelofibrosis, and atypical chronic myeloid leukemia
  * Relapsed or refractory leukemia or MPN that have confirmed JAK mutations and/or positive TSLPR surface staining

    * Testing for JAK mutations and/or confirmed positive flow cytometry surface staining for the thymic stromal lymphopoietin receptor (TSLPR; encoded by CRLF2); eligibility for part C will be contingent upon patients demonstrating overexpression of CRLF2 by flow cytometric methods measured at either JHU or U. Washington flow laboratories (therefore, pre-enrollment samples need to be sent to one of these laboratories after discussion with Dr. Loh) or if the patient has a CLIA lab documented alteration in JAK1 or JAK2, SH2B3, IL7RA, or another gene that would predict sensitivity to JAK inhibition.
* Measurable or evaluable disease (for patients with solid tumors)
* Current disease state is one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* No known active CNS involvement (radiographic or cytologic)

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% (for patients > 16 years old) or Lansky PS 50-100% (for patients ≤ 16 years old)

  * Patients who are unable to walk because of paralysis, but who can actively sit up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance status
* Patients with solid tumors* must meet the following criteria:

  * Peripheral ANC ≥ 1,000/mm^3
  * Platelet count ≥ 100,000/mm^3 (transfusion-independent, defined as > 7 days since prior platelet transfusions)
  * Hemoglobin ≥ 8.0 g/dL (may receive RBC transfusions)

    * Not refractory to to red cell or platelet transfusion
  * ALT ≤ 110 U/L NOTE: *Patients with solid tumors and known bone marrow metastatic disease are eligible for study, but not evaluable for hematologic toxicity. These patients must not be known to be refractory to RBC or platelet transfusions.
* Patients with leukemia or MPNs must meet the following criteria:

  * Platelet count ≥ 20,000/mm^3 (may receive platelet infusions)
  * Hemoglobin ≥ 8.0 g/dL (may receive RBC transfusions)
  * ALT ≤ 225 U/L
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR serum creatinine based on age/gender as follows:

  * ≤ 0.6 mg/dL (for patients 1 to < 2 years old)
  * ≤ 0.8 mg/dL (for patients 2 to < 6 years old)
  * ≤ 1 mg/dL (for patients 6 to < 10 years old)
  * ≤ 1.2 mg/dL (for patients 10 to < 13 years old)
  * ≤ 1.4 mg/dL (for female patients ≥ 13 years old)
  * ≤ 1.5 mg/dL (for male patients 13 to < 16 years old)
  * ≤ 1.7 mg/dL (for male patients ≥ 16 years old)
* Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 times upper limit of normal for age
* Serum albumin ≥ 2 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow crushed or whole tablets

  * Nasogastric or G tube administration is not allowed
* Body surface area ≥ 0.65 m^2 (for patients at dose level -1, 1, and 2)
* No uncontrolled infection, including patients with known active HIV or chronic hepatitis
* No patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

PRIOR CONCURRENT THERAPY:

* Fully recovered from the acute toxic effects of all prior anticancer therapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 months since prior total-body irradiation (TBI), craniospinal radiotherapy, or radiotherapy to ≥ 50% of the pelvis (for patients with solid tumors)
* At least 3 months since prior TBI, craniospinal radiotherapy, or radiotherapy to ≥ 50% of the pelvis (for patients with leukemia)
* At least 3 months since prior stem cell transplantation or rescue without TBI and no evidence of active graft-vs-host disease
* At least 6 weeks since other substantial bone marrow radiation
* At least 3 weeks since prior myelosuppressive therapy (6 weeks for nitrosourea) (for patients with solid tumors)
* At least 2 weeks since prior cytoxic chemotherapy (for patients with leukemia or MPNs)

  * Hydroxyurea may be initiated and continued for up to 24 hours before the start of study treatment
  * Intrathecal cytarabine (Ara-C) is not myelosuppressive chemotherapy
  * Patients with leukemia are permitted to receive intrathecal chemotherapy, including methotrexate or cytarabine, only if this is given at the time of diagnostic lumbar puncture at least 24 hours prior to the start of INCB018424
* At least 2 weeks since prior long-acting hematopoietic growth factor (e.g., Neulasta) or 1 week for a short-acting growth factor

  * For agents that have known adverse events occurring beyond 1 week, this period must be extended beyond the time during which adverse events are known to occur (as discussed with the study chair)
* At least 1 week since prior therapy with a biologic (antineoplastic) agent

  * For agents that have known adverse events occurring beyond 1 week, this period must be extended beyond the time during which adverse events are known to occur (as discussed with the study chair)
* At least 3 half-lives of antibody since prior monoclonal antibody
* No other concurrent investigational drugs
* No other concurrent anticancer agents, including chemotherapy, radiotherapy, immunotherapy, or biologic therapy
* No concurrent systemic steroids (i.e., prednisone > 10 mg)
* No concurrent aspirin > 150 mg/day
* No concurrent medications for myelofibrosis (e.g., hydroxyurea, interferon, thalidomide, busulfan, lenalidomide, or anagrelide)
* No concurrent cyclosporine, tacrolimus, or other agents to prevent graft-vs-host disease after bone marrow transplant or organ rejection after transplant

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2010-09; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose and/or recommended phase II dose | 28 days
Toxicity | 30 days post treatment
Pharmacokinetics | Up to 28 days

SECONDARY OUTCOMES:
Antitumor activity | Up to 30 days post treatment
Toxicity and biologic activity | Day 1 and Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Mignon Loh, MD, Principal Investigator — University of California, San Francisco
Locations (24):
- United States (24):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's Hospital Colorado Center for Cancer and Blood Disorders, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Riley's Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin